CLINICAL TRIAL: NCT01795963
Title: ePREP for Community Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Collaborators: Florida State University (Other); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott R. Braithwaite, Ph.D., Assistant Professor, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2009.2841
Record Dates: First submitted 2013-02-15; First posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Intimate Partner Violence
Keywords: intimate partner violence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Control (Placebo Comparator): Participants in the control condition will view a presentation that teaches inert information about anxiety, depression, and relationships such as definitions, prevalence rates, common problems associated with these conditions and available forms of treatment. This presentation was used initially in Cuckrowicz & Joiner (2007) and has since been shown to be effective as a placebo in two previous ePREP studies (Braithwaite & Fincham, 2007; Braithwaite & Fincham, 2008). This presentation is identical to the ePREP intervention in its set up, the only difference being, there is no information included in this presentation that teaches specific skills or strategies for improving relationships, depression or anxiety.
  Interventions: Behavioral: Placebo Control
- ePREP (Active Comparator): The ePREP intervention teaches individuals how to recognize and combat dynamic risk factors that lead to relationship distress.
  Interventions: Behavioral: ePREP

INTERVENTIONS:
Behavioral: ePREP — The ePREP intervention teaches individuals how to recognize and combat dynamic risk factors that lead to relationship distress. Specifically, it teaches communication techniques and problem-solving skills that help couples to effectively deal with conflict. It also teaches couples how to enhance positive aspects of their relationship by fostering fun and friendship.
  Arms: ePREP
Behavioral: Placebo Control — Participants in the control condition will view a presentation that teaches inert information about anxiety, depression, and relationships such as definitions, prevalence rates, common problems associated with these conditions and available forms of treatment. This presentation was used initially in Cuckrowicz & Joiner (2007) and has since been shown to be effective as a placebo in two previous ePREP studies (Braithwaite & Fincham, 2007; Braithwaite & Fincham, 2008). This presentation is identical to the ePREP intervention in its set up, the only difference being, there is no information included in this presentation that teaches specific skills or strategies for improving relationships, depression or anxiety.
  Arms: Placebo Control

SUMMARY:
The purpose of the present study is to examine the impact of ePREP when it is administered to couples. More specifically, investigators will test whether--compared to placebo controls--participants who receive ePREP will experience better outcomes for relationship relevant variables.

ELIGIBILITY:
Inclusion Criteria:

* Only those who are married or who have been in a committed romantic relationship for six months or longer will be invited to participate.

Exclusion Criteria:

* The only exclusionary criteria were inability to read study questionnaires and unwillingness to access the internet to receive e-mail instructions on weekly homework assignments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Revised Conflict Tactics Scale (CTS-2) | Change across three time-points: baseline, 6-week follow up and 1-year follow up
Communication Patterns Questionnaire (CPQ) | Change across three time-points: baseline, 6-week follow up and 1-year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Braithwaite, Ph.D., Principal Investigator — Brigham Young University
Locations (1):
- Florida State University, Tallahassee, Florida, United States